CLINICAL TRIAL: NCT02219542
Title: Cytokines of Patients After Laparoscopic Colonic Surgery
Brief Title: Cytokines of Patients With Transversus Abdominis Plane Block After Laparoscopic Colonic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wen-fei Tan, Associate proffessor, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20140804
Record Dates: First submitted 2014-08-14; First posted 2014-08-19 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2014-05

CONDITIONS: Laparoscopic Colonic Surgery
Keywords: cytokine Transversus Abdominis Plane Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- a standard general anesthesia (Placebo Comparator): a standard general anesthesia and with transversus abdominis plane block 20 ml 0.9% sodium chloride
  Interventions: Drug: transversus abdominis plane block
- transversus abdominis plane block (Experimental): a standard general anesthesia with transversus abdominis plane block 20 mL 0.25% ropivacaine
  Interventions: Drug: transversus abdominis plane block

INTERVENTIONS:
Drug: transversus abdominis plane block — transversus abdominis plane block with 20 mL saline
  Arms: a standard general anesthesia
Drug: transversus abdominis plane block — transversus abdominis plane block with 20 mL 0.25% ropivacaine
  Arms: transversus abdominis plane block

SUMMARY:
The investigators designed a study to determine whether with combined general-transversus abdominis plane block anesthesia or standard general anaesthetic would provide same level of cytokines in patients undergoing Laparoscopic Colonic Surgery.

DETAILED DESCRIPTION:
The investigators designed a study to determine whether combined general-transversus abdominis plane block anesthesia or standard general anaesthetic would provide same level of cytokine in patients undergoing Laparoscopic Colonic Surgery.

ELIGIBILITY:
Inclusion Criteria:

* •Participants were deemed eligible if they were candidates for spinal anesthesia undergoing Laparoscopic Colonic Surgery

Exclusion Criteria:

* •Existing cognitive impairment as evidenced by Mini-Mental State Examination scores below 24 (of the 30 possible points)

  * A history of neurological and psychiatric diseases including stroke, and psychosis
  * Severe visual or hearing impairment
  * Unwillingness to comply with the protocol or procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The change of cytokine level in plasma samples | just after anesthesia induction ; at the end of the surgery; 24h after surgery
  The blood samples were collected before induction of anesthesia and at the end of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ma, M.D.,PhD, Study Chair — The department of Anesthesiology
Locations (1):
- the First Hospital of China Medical University, Shenyang, Liaoning, China